CLINICAL TRIAL: NCT05323318
Title: Neuropsychological Sequelae as a Risk Factor for Long COVID-19 Fatigue
Brief Title: Neuropsychological Sequelae and Long COVID-19 Fatigue
Acronym: PostCoV2Psy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar Universitario do Algarve (Other)
Collaborators: Universidade do Algarve (Other); Universidade do Porto (Other)
Responsible Party: Principal Investigator, Ligia Pires, Principal Investigator, Centro Hospitalar Universitario do Algarve
Other Study IDs: 141/21
Record Dates: First submitted 2022-04-08; First posted 2022-04-12 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Anxiety Depression; Post Traumatic Stress Disorder; Mental Fatigue; COVID-19; Fatigue Syndrome, Chronic
Keywords: SARS-CoV-2, fatigue, psychological disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mental Fatigue; COVID-19; Fatigue Syndrome, Chronic; Fatigue; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuropsychological Sequelae: Post-COVID-19 symptomatic patients with neuropsychological sequelae
  Interventions: Other: Neuropsychological Sequelae
- Without Neuropsychological Sequelae: Post-COVID-19 symptomatic patients Without neuropsychological sequelae

INTERVENTIONS:
Other: Neuropsychological Sequelae — Neuropsychological Sequelae after SARS-CoV-2 symtomatic infection
  Groups: Neuropsychological Sequelae

SUMMARY:
An association of fatigue with post-viral neuropsychological disturbs has been reported. Among patients hospitalized with COVID-19 there is an increased incidence of anxiety and depression symptoms. In addition, a quarter of patients experience at least mild symptoms of acute post traumatic stress disorder. (Mazza, M. G. et al 2020). The prevalence of chronic fatigue syndrome had a correlation with post-traumatic stress disorder (PTSD) in a study conducted after the outbreak of the COVID-19 in Iran (Silmani et al, 2021), that showed 5.8% of subjects suffering from PTSD after 6 months of SARS-CoV-2 infection onset.

In this Study we propose to use a tool to quantify the degree of physical and psychological fatigue in post-COVID-19 patients, and assess the correlation of fatigue with the neuropsychiatric sequelae in hospitalized and non hospitalized patients.

DETAILED DESCRIPTION:
This study will address the neuropsychiatric sequelae that remain for at least 6 months after SARS-CoV-2 acute infection, as depression, anxiety and/or post-traumatic stress disorder.

The patiensts will be assessed at the post-COVID-19 outpatient clinics of five Portuguese Hospitals. In the first visit (T1) will be collected the demographic characteristics; the medical history; and the screening of acute disease symptoms and severity. In the second visit (T2), the time frame will be at least 6 months after the positive test and no longer than 9 months, a set of structured questionnaires will be provided, including: the Chalder Fatigue Scale, Anxiety and Depression Hospital Scale (HADS), The Posttraumatic Stress Symptoms-14 (PTSS-14) adapted to COVID-19 and the EuroQol 5-Dimensions (EQ-5D).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years;
* Previous COVID-19 at least six months after the diagnosis duly documented in the clinical record;
* Persistent symptoms after cure criteria defined by WHO Symptomatic patients that attend the post-COVID-19 follow-up consultation of the study centres.
* SARS-CoV-2 RNA confirmed by a positive real-time reverse-transcription polymerase chain reaction on a nasopharyngeal swab.
* SARS-CoV-2 antigen confirmed on a nasopharyngeal swab, by a healthcare professional.

Exclusion Criteria:

* Patients with PTSD previous diagnosis
* Severe psychiatric disorders documented in the clinical record
* Patients not able to respond the questionnaire
* Patients who had a concomitant severe neurological disorder
* Clinical and radiological diagnosis of Stroke with sequelae
* Clinical diagnosis of Alzheimer's Disease
* Clinical diagnosis of Parkinson's disease
* Patients with persistent fatigue symptoms in the 6 months before SARS-CoV 2 infection

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in five Portuguese Hospitals, Universitary and district, in which a follow-up post-COVID-19 medical consultation has been implemented
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of fatigue in patients with post-COVID-19 depression and/or anxiety | 6-9 months
  Fatigue will be assessed with the Chalder fatigue scale:
  - Global score (0-33), that also spans two dimensions-physical fatigue (measured by items 1-7) and psychological fatigue (measured by items 8-11). This is a Likert scoring system that allows for means and distributions to be calculated for both the global total as well as the two sub-scales.
  Depression and anxiety will be assessed with the Hospital Anxiety and Depression Scale
  * Depression HADS subscale scoring: Normal 0-7; Boderline abnormal 8-10; Abnormal 11-21
  * Anxiety HADS subscale scoring: Normal 0-7; Borderline 8-10; Abnormal 11-21
Prevalence of fatigue in patients with post-COVID-19 post-traumatic stress disorder | 6-9 months
  Fatigue will be assessed with the Chalder fatigue scale (global and binary score).
  PTSD will be assessed with the Post-Traumatic Stress Syndrome 14 Questions Inventory (PTSS-14) adapted to COVID-19:
  - Positive case between 46-98 points

SECONDARY OUTCOMES:
Impact of post-COVID-19 fatigue in quality of life. | 6-9 months
  Fatigue will be assessed with the Chalder fatigue scale (binary score and global score).
  Quality of live will be assessed by the original EQ-5D questionnaire, that comprises two parts:
  - EQ-5D-3L, health state classification scheme of five items (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each having three alternatives (1= no problems, 2= moderate problems, and 3= severe problems). Calculating a single index score combines these five dimensions.
  The index value of a particular health state thus indicates the preference for being in that health state in relation to death, which has been set equal to 0 and best possible health (eg, no problems on any of the five items) which has been set to 1.0.
  - EQ VAS, a visual analog scale to health state ranging from 0 (worst possible health state) to 100 (best possible health state).
Impact of post-COVID-19 neuropsychological sequelae in quality of life | 6-9 months
  Evaluate if the positive cases for anxiety, depression and/or PTSD have lower quality of live (The tools will be the same of previous outcomes).
Evaluate if neuropsychological are associated with severity of acute COVID-19 | 6-9 months
  Depression and anxiety will be assessed with the Hospital Anxiety and Depression Scale
  * Depression HADS subscale scoring: Normal 0-7; Boderline abnormal 8-10; Abnormal 11-21
  * Anxiety HADS subscale scoring: Normal 0-7; Borderline 8-10; Abnormal 11-21
  Posttraumatic Stress Symptoms-14 instrument, adapted in this protocol for COVID-19 survivors:
  - PTSS 14 scoring > 45 points
  Acute COVID-19 severity will be categorized as mild illness (mild symptoms without the radiographic appearance of pneumonia), pneumonia (having symptoms and the radiographic evidence of pneumonia, with no requirement for supplemental oxygen), severe pneumonia (having pneumonia, including one of the following: respiratory rate > 30 breaths/minute; severe respiratory distress; or SpO2 ≤ 93% on room air at rest), and critical cases (e.g. respiratory failure requiring mechanical ventilation or nasal high flow oxygen, septic shock, other organ failure occurrence or admission into the ICU).

CONTACTS AND LOCATIONS:
Overall Officials: Ligia Pires, MD, Study Chair — Centro Hospitalar Universitario do Algarve; Joana Berger, PHD, Study Director — Universitat Bern; Ligia Pires, MD, Principal Investigator — Centro Hospitalar Universitario do Algarve; Marta Drummond, PHD, Principal Investigator — Universidade do Porto
Locations (6):
- Portugal (6):
  - Hospital Particular de Alvor, Alvor
  - Hospital Professor Doutor Fernando Fonseca (Hff), Amadora
  - Hospital de Faro (Chua), Faro
  - Hospital de Portimao, Portimão
  - Hospital de Sao Sebastiao (Chedv), Santa Maria da Feira
  - Hospital de Vila Franca de Xira (Hvfx), Vila Franca de Xira

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferreira LN, Ferreira PL, Pereira LN, Oppe M. The valuation of the EQ-5D in Portugal. Qual Life Res. 2014 Mar;23(2):413-23. doi: 10.1007/s11136-013-0448-z. Epub 2013 Jun 8. PMID 23748906
- [Background] Jackson C. The Chalder Fatigue Scale (CFQ 11). Occup Med (Lond). 2015 Jan;65(1):86. doi: 10.1093/occmed/kqu168. No abstract available. PMID 25559796
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Rasa S, Nora-Krukle Z, Henning N, Eliassen E, Shikova E, Harrer T, Scheibenbogen C, Murovska M, Prusty BK; European Network on ME/CFS (EUROMENE). Chronic viral infections in myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). J Transl Med. 2018 Oct 1;16(1):268. doi: 10.1186/s12967-018-1644-y. PMID 30285773
- [Result] Simani L, Ramezani M, Darazam IA, Sagharichi M, Aalipour MA, Ghorbani F, Pakdaman H. Prevalence and correlates of chronic fatigue syndrome and post-traumatic stress disorder after the outbreak of the COVID-19. J Neurovirol. 2021 Feb;27(1):154-159. doi: 10.1007/s13365-021-00949-1. Epub 2021 Feb 2. PMID 33528827
- [Result] Mazza MG, De Lorenzo R, Conte C, Poletti S, Vai B, Bollettini I, Melloni EMT, Furlan R, Ciceri F, Rovere-Querini P; COVID-19 BioB Outpatient Clinic Study group; Benedetti F. Anxiety and depression in COVID-19 survivors: Role of inflammatory and clinical predictors. Brain Behav Immun. 2020 Oct;89:594-600. doi: 10.1016/j.bbi.2020.07.037. Epub 2020 Jul 30. PMID 32738287
- [Derived] Pires L, Reis C, Mesquita Facao AR, Moniri A, Marreiros A, Drummond M, Berger-Estilita J. Fatigue and Mental Illness Symptoms in Long COVID: Protocol for a Prospective Cohort Multicenter Observational Study. JMIR Res Protoc. 2024 Jan 19;13:e51820. doi: 10.2196/51820. PMID 38241071